CLINICAL TRIAL: NCT06740565
Title: A Multicenter, Prospective, Randomized Control Study on the Optimal Intervention Approach for High-risk Type B Aortic Dissection
Brief Title: Conventional TEVAR Versus FABULOUS RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Lixin Wang, Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBAD202412
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Type B Aortic Dissection
Keywords: endovascular repair; distal bare stent
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- c-TEVAR (Active Comparator): conventional thoracic endovascular aortic repair
  Interventions: Procedure: thoracic endovascular aortic repair
- Fabulous (Experimental): proximal stent graft combined with distal bare stent
  Interventions: Procedure: thoracic endovascular aortic repair

INTERVENTIONS:
Procedure: thoracic endovascular aortic repair — stent-graft implanted to seal the proximal entry tear of type B aortic dissection

SUMMARY:
For High-risk Type B aortic dissections, a multicenter, prospective, randomized controlled study is conducted to compare the clinical outcomes of conventional proximal endovascular repair (TEVAR) alone versus the Fabulous system which includes a proximal stent graft with a distal bare metal stent implanted. The study aims to determine the optimal intervention method for such population.

DETAILED DESCRIPTION:
Aortic dissection is characterized by its sudden onset, rapid progression, and life-threatening nature, with a natural mortality rate of 25% within 24 hours and 50% within 48 hours. As China's socioeconomic development accelerates and the population continues to age, the incidence of aortic dissection has been rising year by year. According to the China Cardiovascular Health and Disease Report 2022, cardiovascular diseases are now the leading cause of death among urban and rural residents in China. It is estimated that 245 million people in China suffer from hypertension, a major risk factor for aortic dissection. The Sino-RAD study on aortic dissection indicates that, compared to Western countries, China exhibits a "high incidence, early onset" trend, which is related to poor hypertension control. The average age of Chinese aortic dissection patients is 51.8 years, about 10 years younger than in Western countries, which significantly affects life expectancy and imposes a heavy economic burden on healthcare.

Type B aortic dissection refers to dissections originating from the left subclavian artery and beyond. Since 1999, when thoracic endovascular aortic repair (TEVAR) was first introduced internationally, there has been a revolutionary shift in the surgical treatment of B-type aortic dissection, transitioning from highly invasive open surgeries to minimally invasive endovascular treatments. This shift has greatly reduced perioperative mortality and complications. China's treatment of Type B aortic dissection has kept pace with international advancements. Data from the National Center for Cardiovascular Diseases Quality Control shows that from 2017 to 2022, the number of TEVAR surgeries in China increased from 13,709 per year to 24,076 per year, a growth of 75.6%. The number of hospitals performing TEVAR surgeries also increased from 627 to 1,050. However, with the increase in cases, clinical challenges have also emerged.

Type B aortic dissection patients exhibit both common and individual characteristics. Currently, for acute Type B dissections, regardless of subtype, most patients undergo proximal endovascular repair during the subacute phase, while a "watch and wait" strategy is adopted for dissections distal to the descending aorta. This single treatment approach carries potential risks, including inappropriate indications, mistimed interventions, and uncertain prognoses.

Our team has already established a database and imaging library with nearly ten thousand cases. Building on the study of acute complex, non-complex, penetrating ulcers, and intramural hematomas, we are delving deeper into acute high-risk subtypes and localized contrast enhancement of the aortic wall for more refined classifications. For patients with different classifications and at various stages of dissection, such as hyperacute, acute, and subacute phases, it is critical to develop individualized treatment strategies. These strategies may include optimal medical treatment, proximal endovascular repair alone, or a combination of proximal repair and distal petticoat techniques.

Therefore, large-scale clinical research is urgently needed to identify the best intervention timing and methods, based on refined classifications, to establish personalized, stratified diagnosis and treatment strategies for different patients.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 years or older, or non-pregnant females

  * Diagnosed with high-risk Type B aortic dissection with a narrow true lumen (defined as the minimum true lumen diameter being less than 30% of the total vessel diameter) and/or poor radiographic or clinical visceral perfusion (including abnormal blood supply to the liver, kidneys, mesentery, or lower limb ischemia)
  * Deemed suitable for endovascular treatment according to the investigator's judgment
  * Able to understand the purpose of the trial, willing to participate voluntarily and sign the informed consent form, and committed to follow-up visits.

Exclusion Criteria:

* • Subjects with hemodynamic instability or ruptured aortic dissection

  * Subjects who, due to various anatomical factors, are unable to undergo TEVAR alone
  * Subjects with connective tissue diseases, such as Marfan syndrome
  * Subjects in poor general condition, unable to tolerate general anesthesia
  * Subjects allergic to contrast agents, nitinol stent materials, or other stent components
  * Subjects with a life expectancy of less than 12 months
  * Subjects with a history of myocardial infarction or unstable angina within the past 3 months
  * Subjects with a history of TIA or cerebral infarction within the past 3 months
  * Subjects with creatinine levels exceeding 2.5 times the upper normal limit or those currently on dialysis
  * Subjects with severe conditions such as liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
12-Month Positive Aortic Remodeling Rate | 12-month postoperative
  Definition of Positive Aortic Remodeling (meeting at least one of the following criteria). Reduction in the maximum diameter or volume of the false lumen with total aortic diameter or volume growth of less than 5mm or reduction. Increase in the maximum diameter or volume of the true lumen with total aortic diameter or volume growth of less than 5mm or reduction. Reduction in the maximum aortic diameter (with corresponding changes in both true and false lumen diameters).

SECONDARY OUTCOMES:
30-day Composite Major Adverse Events (MAE) Rate | 30-day postoperative
  The incidence of composite major adverse events include cardiac complications, pulmonary complications, renal failure, cerebrovascular complications, limb ischemia, bowel ischemia and spinal cord injury

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol